CLINICAL TRIAL: NCT00110890
Title: An Open-Label, Randomised Study Using Cinacalcet to Improve Achievement of Kidney Disease Outcomes Quality Initiative (K/DOQI) Targets in Patients With ESRD
Brief Title: A Research Study for Patients With End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20030187
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-02

CONDITIONS: End Stage Renal Disease
Keywords: Secondary HyperParaThyroidism (SHPT); Dialysis, End Stage Renal Disease (ESRD); KDOQI, Cinacalcet; Clinical Trial, Amgen
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperparathyroidism, Secondary | interventions — Cinacalcet; Standard of Care

ARMS (2):
- Standard of care (No Intervention): Subjects randomised to the standard care arm are to receive appropriate therapy in accordance with the investigator's practice in an attempt to achieve the K/DOQI PTH, serum calcium, phosphorus, and Ca x P treatment targets.
  Interventions: Other: Standard of care
- Cinacalcet (Other): Treatment with cinacalcet will be initiated at a dose of 30 mg/day. Possible daily doses of cinacalcet are 30, 60, 90, 120, and 180 mg. Dose escalation of cinacalcet may occur based on iPTH values.
  Interventions: Drug: cinacalcet

INTERVENTIONS:
Drug: cinacalcet — Treatment with cinacalcet will be initiated at a dose of 30 mg/day. Possible daily doses of cinacalcet are 30, 60, 90, 120, and 180 mg.
  Arms: Cinacalcet
Other: Standard of care — Subjects randomised to the standard care arm are to receive appropriate therapy in accordance with the investigator's practice in an attempt to achieve the K/DOQI PTH, serum calcium, phosphorus, and Ca x P treatment targets.
  Arms: Standard of care

SUMMARY:
The purpose of this study is to evaluate the ability of a treatment strategy, that includes cinacalcet for the management of secondary hyperparathyroidism, to control parathyroid hormone (PTH) compared with the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients requiring maintenance dialysis (haemodialysis, haemodiafiltration, haemofiltration, or peritoneal dialysis) for at least 1 month
* The mean of 2 iPTH determinations within 21 days before randomization and drawn at least 2 days apart must be greater than or equal to 300 pg/mL (31.8 pmol/L) and less than 800 pg/mL (84.8 pmol/L). If biPTH is determined, the mean levels must be greater than or equal to 150 pg/mL (15.9 pmol/L) and less than 410 pg/mL (43.5 pmol/L)
* The mean of 2 serum calcium determinations (corrected for albumin) drawn on the same day as the PTH determinations must be greater than or equal to 8.4 mg/dL (2.1 mmol/L)

Exclusion Criteria:

* Have an unstable medical condition, defined as having been hospitalised, other than for dialysis vascular access revision, within 30 days before day 1, or otherwise unstable in the judgment of the investigator
* Have had a parathyroidectomy in the 6 months before day 1
* Have received vitamin D therapy for less than 21 days before day 1 or required a change in prescribed vitamin D brand or dose within 21 days before day 1. If subjects are not prescribed vitamin D therapy, they must remain free of vitamin D therapy for the 21 days before day 1.
* Received, within 21 days before day 1 of the dose titration phase, therapy with medications that are predominantly metabolized by the enzyme CYP2D6 and have a narrow therapeutic index (e.g., flecainide, vinblastine, thioridazine, and most tricyclic antidepressants). The tricyclic antidepressant amitriptyline is permitted. - Experienced a myocardial infarction within 3 months prior to day 1
* Are currently enrolled in, or have not yet completed at least 30 days before day 1, other invasive investigational device or investigational drug trials, or are receiving other investigational agents (experimental dialysis machines are acceptable)
* Have a gastrointestinal disorder that may be associated with impaired absorption or orally administered medications or an inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2004-05; Primary Completion 2005-04 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Messa P, Macario F, Yaqoob M, Bouman K, Braun J, von Albertini B, Brink H, Maduell F, Graf H, Frazao JM, Bos WJ, Torregrosa V, Saha H, Reichel H, Wilkie M, Zani VJ, Molemans B, Carter D, Locatelli F. The OPTIMA study: assessing a new cinacalcet (Sensipar/Mimpara) treatment algorithm for secondary hyperparathyroidism. Clin J Am Soc Nephrol. 2008 Jan;3(1):36-45. doi: 10.2215/CJN.03591006. PMID 18178780
- [Result] Wilkie M, Pontoriero G, Macario F, Yaqoob M, Bouman K, Braun J, von Albertini B, Brink H, Maduell F, Graf H, Frazao JM, Bos WJ, Torregrosa V, Saha H, Reichel H, Zani VJ, Carter D, Messa P. Impact of vitamin D dose on biochemical parameters in patients with secondary hyperparathyroidism receiving cinacalcet. Nephron Clin Pract. 2009;112(1):c41-50. doi: 10.1159/000212102. Epub 2009 Apr 10. PMID 19365139
- [Derived] Frazao JM, Braun J, Messa P, Dehmel B, Mattin C, Wilkie M. Is serum phosphorus control related to parathyroid hormone control in dialysis patients with secondary hyperparathyroidism? BMC Nephrol. 2012 Aug 3;13:76. doi: 10.1186/1471-2369-13-76. PMID 22863242
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 28 May 2004 through 12 November 2004
Groups:
- Cinacalcet: Treatment with cinacalcet will be initiated at a dose of 30 mg/day. Possible daily doses of cinacalcet are 30, 60, 90, 120, and 180 mg. Dose escalation of cinacalcet may occur based on intact parathyroid hormone (iPTH) values.
- Standard of Care: Subjects randomised to the standard care arm are to receive appropriate therapy in accordance with the investigator's practice in an attempt to achieve the Kidney Disease Outcomes Quality Initiative (K/DOQI) parathyroid hormone (PTH), serum calcium, phosphorus, and Ca x P treatment targets.
Period: Overall Study
Arm/Group | Cinacalcet | Standard of Care
Started | 368 | 184
End of Dose Optimization Phase | 316 (Weeks 1 to 16) | 170 (Weeks 1 to 16)
End of Efficacy Assessment Phase | 280 (Weeks 17 to 23) | 150 (Weeks 17 to 23)
Completed | 7 (Follow-up Phase) | 5 (Follow-up Phase)
Not Completed | 361 | 179
Not completed — Adverse Event | 30 | 7
Not completed — Death | 16 | 9
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 4 | 5
Not completed — Withdrawal by Subject | 17 | 5
Not completed — Protocol Deviation | 1 | 0
Not completed — Noncompliance | 10 | 0
Not completed — Kidney Transplant | 16 | 12
Not completed — Invest. Product Commercially Available | 217 | 110
Not completed — Other | 34 | 23
Not completed — Ineligibility determined | 3 | 0
Not completed — Requirement for alternative therapy | 0 | 1
Not completed — Disease progression | 0 | 1
Not completed — Parathyroidectomy | 0 | 1
Not completed — Did not enter follow-up phase | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinacalcet | Standard of Care | Total
Number analyzed (Participants) | 368 | 184 | 552
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (14.5) | 58.3 (14.5) | 58.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 67 | 211
  Male | 224 | 117 | 341
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 349 | 172 | 521
  Black | 9 | 7 | 16
  Other | 5 | 5 | 10
  Unknown | 5 | 0 | 5
Baseline Strata [Number; unit: Participants]
  Vitamin D prescribed and Ca x P ≤ 55 mg^2/dL^2 | 158 | 79 | 237
  Vitamin D prescribed and Ca x P > 55 mg^2/dL^2 | 94 | 47 | 141
  Vitamin D not prescribed and Ca x P ≤ 55 mg^2/dL^2 | 69 | 34 | 103
  Vitamin D not prescribed and Ca x P > 55 mg^2/dL^2 | 47 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mean PTH ≤ 300 pg/mL
Description: Number of participants with mean parathyroid hormone (PTH) ≤ 300 pg/mL during the efficacy assessment phase
Time Frame: Efficacy Assessment Phase (weeks 17 to 23)
Population: Full Analysis Set, composed of all randomized participants with imputation using modified last value carried forward (mLVCF)
Measure: Number; unit: Participants
Arm/Group | Cinacalcet | Standard of Care
Number analyzed (Participants) | 368 | 184
Participants | 262 | 41
Statistical Analysis 1: Comparison: Cinacalcet vs Standard of Care; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2; Odds Ratio (OR) = 8.74, 95% CI [5.72 to 13.36] — Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2

2. Secondary Outcome: Number of Participants With Mean Ca x P < 55 mg^2/dL^2 and iPTH ≤ 300 pg/mL
Description: Number of participants with mean calcium x phosphorus (Ca x P) < 55 mg^2/dL^2 and intact parathyroid hormone (iPTH) ≤ 300 pg/mL during the efficacy assessment phase
Time Frame: Efficacy Assesment Phase (weeks 17-23)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cinacalcet | Standard of Care
Number analyzed (Participants) | 368 | 184
Participants | 217 | 29
Statistical Analysis 1: Comparison: Cinacalcet vs Standard of Care; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2; Odds Ratio (OR) = 8.74, 95% CI [5.38 to 14.19] — Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2

3. Secondary Outcome: Number of Participants With Mean Ca x P < 55 mg^2/dL^2
Description: Number of participants with mean calcium x phosphorus (Ca x P) < 55 mg^2/dL^2 during the efficacy assessment phase
Time Frame: Efficacy Assessment Phase (weeks 17 to 23)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cinacalcet | Standard of Care
Number analyzed (Participants) | 368 | 184
Participants | 282 | 106
Statistical Analysis 1: Comparison: Cinacalcet vs Standard of Care; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2; Odds Ratio (OR) = 3.11, 95% CI [2.00 to 4.84] — Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2

4. Secondary Outcome: Number of Participants With Mean Serum Ca < 9.5 mg/dL
Description: Number of participants with mean serum calcium (Ca) < 9.5 mg/dL during the efficacy assessment phase
Time Frame: Efficacy Assessment Phase (weeks 17-23)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cinacalcet | Standard of Care
Number analyzed (Participants) | 368 | 184
Participants | 281 | 61
Statistical Analysis 1: Comparison: Cinacalcet vs Standard of Care; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2; Odds Ratio (OR) = 6.93, 95% CI [4.65 to 10.34] — Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2

5. Secondary Outcome: Number of Participants With Mean Serum P < 5.5 mg/dL
Description: Number of participants with mean serum phosphorus (P) < 5.5 mg/dL during the efficacy assessment phase
Time Frame: Efficacy Assessment Phase (weeks 17 to 23)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cinacalcet | Standard of Care
Number analyzed (Participants) | 368 | 184
Participants | 231 | 92
Statistical Analysis 1: Comparison: Cinacalcet vs Standard of Care; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2; Odds Ratio (OR) = 1.88, 95% CI [1.26 to 2.81] — Adjusted for four baseline strata defined by vitamin D prescribed and calcium x phosphorus ≤ 55 mg^2/dL^2

ADVERSE EVENTS:
Time Frame: 23 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Standard Care | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 31/182 | 83/365
Other Adverse Events (participants affected / at risk) | 31/182 | 173/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care (N=182) | Cinacalcet (N=365)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 3
Arrhythmia (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac asthma (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Catheter related complication (General disorders) | 0 | 2
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Sudden cardiac death (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 2
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchitis acute (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 2
Catheter related infection (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 0 | 1
Clostridium bacteraemia (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 2
Graft infection (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Perianal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 1
Renal cyst infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 3
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Device failure (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 2
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 2
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem ischaemia (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Catheter placement (Surgical and medical procedures) | 1 | 1
Nephrectomy (Surgical and medical procedures) | 1 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral circulatory failure (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Phlebothrombosis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care (N=182) | Cinacalcet (N=365)
Diarrhoea (Gastrointestinal disorders) | 12 | 47
Nausea (Gastrointestinal disorders) | 6 | 115
Vomiting (Gastrointestinal disorders) | 12 | 87
Nasopharyngitis (Infections and infestations) | 6 | 27
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.